CLINICAL TRIAL: NCT04778202
Title: Diagnostic and Prognostic Value of MicroRNA as a Potential Biomarker in Breast Cancer Patients in Correlation to Radiological Findings.
Brief Title: Diagnostic and Prognostic Value of MicroRNA in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, asmaa saleh abdelghfour, demonstrator, Assiut University
Other Study IDs: MicroRNA in breast cancer
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample by veinpuncture prosedure into EDITA tubes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- first group (control group): 25 normal health control women apparently healthy. blood samples will be obtained after getting informed consent
  Interventions: Diagnostic Test: blood sample collection
- Second group (breast cancer patient group): 25 female patients referred to radiology departement at South Egypt Cancer Institute or Assiut University Hospital diagnosed as breast cancer patients as evidenced by clinical examination , mammography and histopathology
  Interventions: Diagnostic Test: blood sample collection

INTERVENTIONS:
Diagnostic Test: blood sample collection — blood sample collection by venipuncture four both groups and MRI for breast cancr patient group

SUMMARY:
The aim of this study is to evaluate the role of miRNA 125a -5p and miRNA143-3p as a non invasive biomarker in diagnosis of breast cancer and the relationship between MiRNA expression and histopathological features as tumor stage ,grade ,molecular subtypes. Also trying to correlate the results with MRI radiological findings which may help in better selection of treatment protocols.

DETAILED DESCRIPTION:
Breast cancer ( BC) is the most commonly diagnosed cancer in women worldwide. The incidence and mortality rates for female breast cancer far exceeded those for other cancers . Although the incidence rate of breast cancer has risen, the mortality rates have steadily fallen due to early diagnosis and better treatments . Early detection of breast cancer often leads to better outcomes. According to Cancer Australia's National Cancer Control Indicators, the relative survival for females diagnosed with early-stage breast cancers at diagnosis was much higher than that for those with advanced breast diagnosis.

Despite the improvement in diagnosis and treatment,approximately 20% of BC patients will develop metastasis.This setting is considered an incurable disease that often occurs due to either resistance to therapy or diagnosis at advanced stages . In this scenario, although 44% of the patients are diagnosed at stage I (AJCC cancer staging) with 5-year survival rates of 100%, 5% of patients are diagnosed at stage IV with 5-year survival rates of approximately 26% .

The small percentage of women diagnosed at advanced stage of the disease gives evidence that mammography represents the best available screening option for breast cancer .

However, more accurate and meaningful early-diagnosis methods together with image techniques would improve BC survival rates.

MicroRNAs (MiRNAs) are short endogenous noncoding RNA molecules of 19-25 nt that have important gene regulatory roles at post-transcriptional level [8, 9]. They pair with messenger RNAs (mRNAs) of protein-coding genes and depending on complementarity, leading to mRNa translational repression or degradation . They regulate 30% of transcripts and contain 3% of the human genome .

In the past few years, miRNAs were established as relevant molecular components of cells in normal or malignant processes.. Particularly, miRNAs have been demonstrated to have an important role in cancer biology through post transcriptional editing of target messenger RNAs expression involved in tumor growth, invasion, metastasis or immune escape .

In addition, several tumor-associated miRNA profiles have been proposed and investigated as biomarkers for diagnosis, survival, response to treatment or tumor subclassification.

The development of early diagnostic tools is of most interest to the clinics since early diagnosis is associated with better prognosis.

In this context, miRNAs have been demonstrated to be good early diagnostic biomarkers in several types of cancer including BC, among others.

One of the main advantages of circulating miRNAs is their high stability in body fluids , which is the main reason for them to be used in cancer diagnosis or prognosis.

Moreover, the assessment of circulating miRNAs can be carried out with simple, lowcost and quick assays.

These characteristics highlight the value of miRNAs as non-invasive biomarkers. Indeed, several miRNAs have been found to be differentially expressed in blood, plasma or serum from healthy donors compared with BC patients, supporting their use as noninvasive, early-stage diagnosis biomarkers.

Growing evidences revealed that imaging techniques are associated with some limitations such as expensive. Hence, it seems that utilization of improvement imaging techniques and biochemistry biomarkers could overcome the limitations associated with imaging techniques. Beside utilization of imaging techniques, identification of new biomarkers in patients with breast cancer has provided an interesting landscape .

So studies have identified different circulating miRNAs as new biomarkers for BC detection; Moreover, they have not been assessed in conjunction with diagnostic imaging, which is used for quantifying the extent of the disease and provides information related to tumour aggressiveness representing an obligatory step for treatment planning. The use of diagnostic imaging to extract quantitative parameters related to the morphology, metabolism and functionality of tumours, as well as to correlate specific imaging parameters with molecular biomarkers, is an emerging research topic

ELIGIBILITY:
Inclusion Criteria:

1. control group of normal healthy individuals who don't have tumors in other organs.
2. breast cancer group Patients with confirmed breast cancer who didn't receive radiotherapy ,chemotherapy ,hormonal therapy or surgical treatment.

Exclusion Criteria:

1. Patients refuse to be part of study and undergo examination .
2. All patients with breast cancer that had received chemotherapy, radiotherapy , ,hormonal or surgical treatment.
3. History of benign or malignant tumors in other organs

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: females 18 years old or above
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
assessment of the value of MiRNA in diagnosis and prognosis of breast cancer patients | 18-24 month
  To evaluate diagnostic and prognostic role of MiRNA 125a-5p and 143-3p as a non invasive biomarker in breast cancer
correlat MiRNA expression with MRI findings for better selection of treatment plan and out come | 18-24 months
  Also trying to correlate the results with MRI radiological findings which may help in better selection of treatment protocols.

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593